CLINICAL TRIAL: NCT06804551
Title: A Single-center, Prospective, Double-blind, Randomized Controlled Trial Evaluating Iovera° Lumbar Medial Branch Cryoneurolysis Versus Radiofrequency Ablation for the Treatment of Facet-mediated Chronic Low Back Pain
Brief Title: Cryoneurolysis Versus Radiofrequency Ablation for the Treatment of Chronic Low Back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY00160986
Record Dates: First submitted 2025-01-07; First posted 2025-02-03 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Chronic Low-back Pain
Keywords: iovera; radiofrequency ablation; medial branch block; chronic low back pain; cryoneurolysis
MeSH Terms: interventions — Radiofrequency Ablation

STUDY DESIGN:
Intervention Model Description: Prospective, double-blind, randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, investigators, clinician, assessors and biostatistician are blinded to the treatment allocation through use of physical blinds to the intervention being administered and coded participant ID's.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- iovera system (Active Comparator): Uses liquid nitrous oxide contained within the device and a closed-end needle to create a precise zone of cold to denature the target medial branch nerve supplying the facet joint by Wallerian degeneration (second degree axonotmesis) preserving the epineurium, perineurium, and endoneurium.
  Interventions: Device: iovera system
- Radiofrequency ablation (Active Comparator): Utilizes radiofrequency energy to heat and denature the target medial branch nerve supplying the facet joint.
  Interventions: Device: Radiofrequency ablation alone

INTERVENTIONS:
Device: iovera system — Reusable, portable Handpiece, along with single patient use sterile Smart Tips (i.e., cryoprobes) and disposable nitrous oxide (N2O) cartridges. The iovera° system produces the desired effect through initiation of a cooling cycle. Each cooling cycle is initiated by fully inserting the Smart Tip into the selected procedure site and activating the cryogen flow. The Smart Tip needles are made of stainless steel and have a closed tip, fully enclosing the cryogen. The STT21180STIM Smart Tip will be used in this study.
  Other Names: Cryoneurolysis
  Arms: iovera system
Device: Radiofrequency ablation alone — An electrode at the tip of the needle sends radio waves that lesion the nerve bundles.
  Other Names: Ablation
  Arms: Radiofrequency ablation

SUMMARY:
Low back pain (LBP) is the leading cause of disability worldwide. Currently available treatment options for treating low back facet joint pain include acupuncture, pain medications, psychotherapy, anti-inflammatory steroid injections into the joints, exercise, physical therapy, rest, chiropractic treatments, surgery, and radiofrequency ablation (RFA). RFA uses radio waves to target and burn the nerves that send the pain signals to the participant's brain. The purpose of this study is to compare the standard treatment of RFA to a newer therapy called iovera°. The iovera° system is a newer procedure for nerve pain that freezes the targeted nerves leading to a temporary block of the nerve without causing any permanent damage to the nerve. With the nerve blocked, pain is immediately relieved. The nerve reconnects over time and goes back to working exactly as it did before the procedure. The investigators want to see if iovera° therapy is effective in treating people with facet joint-mediated chronic low back pain (CLBP).

If the participant decide to participate in the study, the investigators will ask the participant to undergo either an RFA or iovera° procedure to treat the participant's CLBP. After the procedure, the investigators will ask the participant to complete surveys to track the participant's response to the procedure at 15 time points over a 1-year period. These time points consist of phone calls and online surveys.

DETAILED DESCRIPTION:
Potential subjects will be screened within 30 days prior to the iovera° treatment. After the Informed Consent Form (ICF) is signed, demographic information (including the Pain Catastrophizing Scale (PCS), Oswestry Disability index (ODI), and Patient Health Questionnaire (PHQ-9)), medical and surgical history, concomitant medications/concurrent procedures information, and vital signs will be collected. An assessment of the intended treatment areas will be conducted. Subjects will assess the pain in their low back region using a Numeric Rating Scale (NRS) and health-related quality of life (EQ-5D-5L) at the screening visit. When screening test results are received and the subject is deemed eligible for the study, the subject will be notified that he or she is enrolled in the study and will receive study procedure.

Study Procedures are Radiofrequency ablation (RFA) and the iovera° system. The site investigators will be trained to perform RFA and to use the iovera° device and a single unblinded research team member will administer the iovera° procedure. The procedure administering investigator(s) will not perform any of the study-specific assessments.

Post-treatment:

After the study procedure, subjects will be instructed to take their prescribed pain medications (i.e., opioid and non-opioid) as needed in response to their pain experience and record their pain score before taking their medication.

Subjects must be instructed to report any adverse device effects and adverse events (AEs) to the Investigator from the time the ICF is signed through Day 360 (±7 days). Safety will be assessed while subjects are in the facility. The total duration of study follow-up will 360 days (± 7 days). Adverse device effects, serious adverse device effects, adverse events, and serious adverse events will be recorded from the time the ICF is signed through Day 360 (± 7 days). Any concomitant medications used to treat AEs through postsurgical Day 360 (± 7 days) will also be recorded.

ELIGIBILITY:
Inclusion Criteria: Subjects must meet all the following inclusion criteria to be eligible for participation.

* Subjects at least 18 years of age at Screening
* Chronic low back pain (≥ 3 months)
* Successful trial of two diagnostic medial branch blocks
* Failure of at least three months of conservative non-operative therapy (e.g., physical therapy, chiropractic care, sleep hygiene, weight loss, spinal injections, NSAIDs, physician-directed exercise program or other appropriate pain medicine)
* Able to provide informed consent, adhere to the study visit schedule, and complete all study assessments

Exclusion Criteria: Subjects who meet any of the following exclusion criteria will not be eligible for participation in this study.

* Active workers' compensation, personal injury, Social Security disability insurance (SSDI), or other litigation/compensation related to the spine
* Infection in the back or open wounds in the back
* Cancer
* Fractures in the back
* Pain shooting down the leg
* Pain when walking up/downhill
* Any back surgery or metal objects in the back
* Any implants of any kind in the body
* Currently pregnant, nursing, or planning to become pregnant during the study
* Blood clots
* History of RFA treatment in back
* Drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-07 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Confirm the feasibility of a double-blinded protocol | After the last End of Study Visit
  At the end of the study, all of the study team members will fill out a structured questionnaire to determine the feasibility. This questionnaire will include the following:
  1. Considering you role in this study, is it feasible to continue to an efficacy Randomized Control Trial applying the same protocols and procedures used in the current pilot study without modifications?
  2. If not, considering you role in this study, is it feasible to continue to an efficacy Randomized Control Trial applying modifications to the protocols and procedures used in the current pilot study?
  As the aim of this pilot study is not to assess effectiveness or efficacy, formal hypothesis testing will not be determined.

SECONDARY OUTCOMES:
Current pain intensity scores in the low back region | Screening, pretreatment, once daily during Days 1-6, Day 7 ± 2, Day 15 ± 3 days, Day 30 ± 5, Day 60 ± 5, Day 90 ± 5, Day 120 ± 5, Day 150 ± 5, Day 180 ± 5, Day 210 ± 7, Day 240 ± 7, Day 270 ± 7, Day 300 ± 7, Day 330 ± 7, Day 360 ± 7.
  Current pain: subjects will be asked "How much pain are you experiencing in your low back right now?"
  This outcome measures current pain intensity (i.e., pain "right now" in the low back region) using an 11-point Numeric Rating Scale (NRS) instrument in which 0 =no pain and 10 =the worst pain imaginable.
Daily pain intensity scores in the low back region | Screening, pretreatment, once daily during Days 1-6, Day 7 ± 2, Day 15 ± 3 days, Day 30 ± 5, Day 60 ± 5, Day 90 ± 5, Day 120 ± 5, Day 150 ± 5, Day 180 ± 5, Day 210 ± 7, Day 240 ± 7, Day 270 ± 7, Day 300 ± 7, Day 330 ± 7, Day 360 ± 7.
  Daily pain: subjects will be asked "What was your worst pain in the past 24 hours in your low back?" and "What was your average pain in the last 24 hours in your low back?"
  This outcome measures daily pain intensity (i.e., average / worst pain over the past 24 hours in the low back region) using an 11-point Numeric Rating Scale (NRS) instrument in which 0 =no pain and 10 =the worst pain imaginable.
Concomitant medication use | Screening, once daily during Days 1-6, Day 7 ± 2, Day 15 ± 3 days, Day 30 ± 5, Day 60 ± 5, Day 90 ± 5, Day 120 ± 5, Day 150 ± 5, Day 180 ± 5, Day 210 ± 7, Day 240 ± 7, Day 270 ± 7, Day 300 ± 7, Day 330 ± 7, Day 360 ± 7.
  This outcome will record the types, doses and frequencies for concomitant medications used (including opioids and analgesics).
Functional disability | Screening, Day 30 ± 5, Day 60 ± 5, Day 90 ± 5, Day 120 ± 5, Day 150 ± 5, Day 180 ± 5, Day 210 ± 7, Day 240 ± 7, Day 270 ± 7, Day 300 ± 7, Day 330 ± 7, Day 360 ± 7.
  This outcome will be measured using the Oswestry Disability Index (ODI) Questionnaire; the ODI ranges from 0 to 100. A higher score on the ODI indicates a more severe disability caused by low back pain.
Patients' global impression of change | Day 30 ± 5, Day 60 ± 5, Day 90 ± 5, Day 120 ± 5, Day 150 ± 5, Day 180 ± 5, Day 210 ± 7, Day 240 ± 7, Day 270 ± 7, Day 300 ± 7, Day 330 ± 7, Day 360 ± 7.
  This outcome will be measured using the 7-point Patient Global Impression of Change scale regarding change:
  Participants will be asked:
  "Since beginning treatment at this clinic, how would you describe the change (if any) in activity libations, symptoms, emotions, and overall quality of life, related to your painful condition? (circle one number below):
  1. No change (or condition has gotten worse)
  2. Almost the same, hardly any change at all
  3. A little better, but no noticeable change
  4. Somewhat better, but the change has not made any real difference
  5. Moderately better and a slight but noticeable change
  6. Better, and definite improvement that has made a real and worthwhile difference
  7. A great deal better, and a considerable improvement that has made all the difference"
Patients' impression of change | Day 30 ± 5, Day 60 ± 5, Day 90 ± 5, Day 120 ± 5, Day 150 ± 5, Day 180 ± 5, Day 210 ± 7, Day 240 ± 7, Day 270 ± 7, Day 300 ± 7, Day 330 ± 7, Day 360 ± 7.
  This outcome will be measured using the additional 0-10 point question regarding change:
  Participants will be asked:
  "Please circle the number (0-10) that matches your degree of change since the beginning of care at this study: 0 being much better 5 being no change 10 being much worse"
Patient satisfaction with pain management | Day 30 ± 5, Day 60 ± 5, Day 90 ± 5, Day 120 ± 5, Day 150 ± 5, Day 180 ± 5, Day 210 ± 7, Day 240 ± 7, Day 270 ± 7, Day 300 ± 7, Day 330 ± 7, Day 360 ± 7.
  This outcome will be measured with the following scale:
  "Please circle the number below that best describes your overall satisfaction with your pain management. (Select one number only)
  1. Extremely dissatisfied
  2. Dissatisfied
  3. Neither satisfied nor dissatisfied
  4. Satisfied
  5. Extremely satisfied"
Health Related Quality of Life | Screening, Day 90 ± 5, Day 180 ± 5, Day 270 ± 7, Day 360 ± 7.
  This outcome will be measured with the EuroQol (EQ-5D-5L) Validity in Assessing the Quality of Life Questionnaire, a 5 question questionnaire regarding quality of life, with higher values being better health and lower values being worse health).
Pain Catastrophizing | Screening, Day 90 ± 5, Day 180 ± 5, Day 270 ± 7, Day 360 ± 7.
  This outcome will be measured with the Pain Catastrophizing Scale with 0 being not al all to 4 being all the time.
Adverse device effects | This outcome will be recorded from the time the study ICF is signed through Day 360± 7 days.
  The study team will keep a record a descriptive list of any adverse effects that occur pertaining to the device used in the study.
Adverse Events (AE's) | This outcome will be recorded from the time the study ICF is signed through Day 360± 7 days.
  The study team will keep a record of any adverse effects that occur pertaining the participants enrolled in the study. CTCAE v5.0 will be used to classify AE's.
serious adverse events (SAEs) | This outcome will be recorded from the time the study ICF is signed through Day 360± 7 days.
  The study team will keep a record of any serious adverse events that occur pertaining the participants enrolled in the study. CTCAE v5.0 will be used to classify SAE's.

CONTACTS AND LOCATIONS:
Overall Officials: Neil A Segal, MS, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Winston P, Mills PB, Reebye R, Vincent D. Cryoneurotomy as a Percutaneous Mini-invasive Therapy for the Treatment of the Spastic Limb: Case Presentation, Review of the Literature, and Proposed Approach for Use. Arch Rehabil Res Clin Transl. 2019 Oct 17;1(3-4):100030. doi: 10.1016/j.arrct.2019.100030. eCollection 2019 Dec. PMID 33543059
- [Background] Tetzlaff W, Bisby MA. Neurofilament elongation into regenerating facial nerve axons. Neuroscience. 1989;29(3):659-66. doi: 10.1016/0306-4522(89)90138-3. PMID 2500618
- [Background] Starr JB, Gold L, McCormick Z, Suri P, Friedly J. Trends in lumbar radiofrequency ablation utilization from 2007 to 2016. Spine J. 2019 Jun;19(6):1019-1028. doi: 10.1016/j.spinee.2019.01.001. Epub 2019 Jan 10. PMID 30639589
- [Background] Shaffer JP, Williams VB, Shin SS. Cryoneurolysis for Digital Neuralgia in Professional Baseball Players: A Case Series. Orthop J Sports Med. 2022 May 12;10(5):23259671221096095. doi: 10.1177/23259671221096095. eCollection 2022 May. PMID 35601731
- [Background] Sayed D, Grider J, Strand N, Hagedorn JM, Falowski S, Lam CM, Tieppo Francio V, Beall DP, Tomycz ND, Davanzo JR, Aiyer R, Lee DW, Kalia H, Sheen S, Malinowski MN, Verdolin M, Vodapally S, Carayannopoulos A, Jain S, Azeem N, Tolba R, Chang Chien GC, Ghosh P, Mazzola AJ, Amirdelfan K, Chakravarthy K, Petersen E, Schatman ME, Deer T. The American Society of Pain and Neuroscience (ASPN) Evidence-Based Clinical Guideline of Interventional Treatments for Low Back Pain. J Pain Res. 2022 Dec 6;15:3729-3832. doi: 10.2147/JPR.S386879. eCollection 2022. PMID 36510616
- [Background] Rubin DI. Epidemiology and risk factors for spine pain. Neurol Clin. 2007 May;25(2):353-71. doi: 10.1016/j.ncl.2007.01.004. PMID 17445733
- [Background] Rubenstein J, Harvey AW, Vincent D, Winston P. Cryoneurotomy to Reduce Spasticity and Improve Range of Motion in Spastic Flexed Elbow: A Visual Vignette. Am J Phys Med Rehabil. 2021 May 1;100(5):e65. doi: 10.1097/PHM.0000000000001624. No abstract available. PMID 33105153
- [Background] Radnovich R, Scott D, Patel AT, Olson R, Dasa V, Segal N, Lane NE, Shrock K, Naranjo J, Darr K, Surowitz R, Choo J, Valadie A, Harrell R, Wei N, Metyas S. Cryoneurolysis to treat the pain and symptoms of knee osteoarthritis: a multicenter, randomized, double-blind, sham-controlled trial. Osteoarthritis Cartilage. 2017 Aug;25(8):1247-1256. doi: 10.1016/j.joca.2017.03.006. Epub 2017 Mar 20. PMID 28336454
- [Background] Perolat R, Kastler A, Nicot B, Pellat JM, Tahon F, Attye A, Heck O, Boubagra K, Grand S, Krainik A. Facet joint syndrome: from diagnosis to interventional management. Insights Imaging. 2018 Oct;9(5):773-789. doi: 10.1007/s13244-018-0638-x. Epub 2018 Aug 8. PMID 30090998
- [Background] Mehta CR, Pocock SJ. Adaptive increase in sample size when interim results are promising: a practical guide with examples. Stat Med. 2011 Dec 10;30(28):3267-84. doi: 10.1002/sim.4102. Epub 2010 Nov 30. PMID 22105690
- [Background] Manchikanti L, Singh V, Datta S, Cohen SP, Hirsch JA; American Society of Interventional Pain Physicians. Comprehensive review of epidemiology, scope, and impact of spinal pain. Pain Physician. 2009 Jul-Aug;12(4):E35-70. PMID 19668291
- [Background] Manchikanti L, Kaye AD, Soin A, Albers SL, Beall D, Latchaw R, Sanapati MR, Shah S, Atluri S, Abd-Elsayed A, Abdi S, Aydin S, Bakshi S, Boswell MV, Buenaventura R, Cabaret J, Calodney AK, Candido KD, Christo PJ, Cintron L, Diwan S, Gharibo C, Grider J, Gupta M, Haney B, Harned ME, Helm Ii S, Jameson J, Jha S, Kaye AM, Knezevic NN, Kosanovic R, Manchikanti MV, Navani A, Racz G, Pampati V, Pasupuleti R, Philip C, Rajput K, Sehgal N, Sudarshan G, Vanaparthy R, Wargo BW, Hirsch JA. Comprehensive Evidence-Based Guidelines for Facet Joint Interventions in the Management of Chronic Spinal Pain: American Society of Interventional Pain Physicians (ASIPP) Guidelines Facet Joint Interventions 2020 Guidelines. Pain Physician. 2020 May;23(3S):S1-S127. PMID 32503359
- [Background] Katz JN. Lumbar disc disorders and low-back pain: socioeconomic factors and consequences. J Bone Joint Surg Am. 2006 Apr;88 Suppl 2:21-4. doi: 10.2106/JBJS.E.01273. PMID 16595438
- [Background] Guirguis M, Hakkinen I, Amiri JP, Posas J. Cryotherapy. Deer's Treatment of Pain: Springer; 2019:283-289.
- [Background] Evans PJ, Lloyd JW, Green CJ. Cryoanalgesia: the response to alterations in freeze cycle and temperature. Br J Anaesth. 1981 Nov;53(11):1121-7. doi: 10.1093/bja/53.11.1121. PMID 7326160
- [Background] Dasa V, Lensing G, Parsons M, Harris J, Volaufova J, Bliss R. Percutaneous freezing of sensory nerves prior to total knee arthroplasty. Knee. 2016 Jun;23(3):523-8. doi: 10.1016/j.knee.2016.01.011. Epub 2016 Feb 10. PMID 26875052
- [Background] Cohen SP, Raja SN. Pathogenesis, diagnosis, and treatment of lumbar zygapophysial (facet) joint pain. Anesthesiology. 2007 Mar;106(3):591-614. doi: 10.1097/00000542-200703000-00024. PMID 17325518
- [Background] Cohen SP, Bhaskar A, Bhatia A, Buvanendran A, Deer T, Garg S, Hooten WM, Hurley RW, Kennedy DJ, McLean BC, Moon JY, Narouze S, Pangarkar S, Provenzano DA, Rauck R, Sitzman BT, Smuck M, van Zundert J, Vorenkamp K, Wallace MS, Zhao Z. Consensus practice guidelines on interventions for lumbar facet joint pain from a multispecialty, international working group. Reg Anesth Pain Med. 2020 Jun;45(6):424-467. doi: 10.1136/rapm-2019-101243. Epub 2020 Apr 3. PMID 32245841
- [Background] Chou R, Atlas SJ, Stanos SP, Rosenquist RW. Nonsurgical interventional therapies for low back pain: a review of the evidence for an American Pain Society clinical practice guideline. Spine (Phila Pa 1976). 2009 May 1;34(10):1078-93. doi: 10.1097/BRS.0b013e3181a103b1. PMID 19363456
- [Background] Cassidy JD, Carroll LJ, Cote P. The Saskatchewan health and back pain survey. The prevalence of low back pain and related disability in Saskatchewan adults. Spine (Phila Pa 1976). 1998 Sep 1;23(17):1860-6; discussion 1867. doi: 10.1097/00007632-199809010-00012. PMID 9762743
- [Background] Birkenmaier C, Veihelmann A, Trouillier H, Hausdorf J, Devens C, Wegener B, Jansson V, von Schulze Pellengahr C. Percutaneous cryodenervation of lumbar facet joints: a prospective clinical trial. Int Orthop. 2007 Aug;31(4):525-30. doi: 10.1007/s00264-006-0208-6. Epub 2006 Aug 23. PMID 16927087
- [Background] Barnard D. The effects of extreme cold on sensory nerves. Ann R Coll Surg Engl. 1980 May;62(3):180-7. PMID 7396346